CLINICAL TRIAL: NCT03531632
Title: A Phase 1b/2, Open Label, Dose Escalation Study of MGD007, a Humanized gpA33 × CD3 DART® Protein in Combination With MGA012, an Anti-PD-1 Antibody, in Patients With Relapsed or Refractory Metastatic Colorectal Carcinoma
Brief Title: MGD007 Combined With MGA012 in Relapsed/Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD007-02
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGD007 + MGA012 (Experimental): MGD007 is a gpA33 x CD3 bi-specific DART antibody; MGA012 is an anti-PD-1 monoclonal antibody.
  Interventions: Biological: MGD007 + MGA012

INTERVENTIONS:
Biological: MGD007 + MGA012 — MGD007 and MGA012 are administered by IV infusion.
  Other Names: MGA012 also known as INCMGA00012

SUMMARY:
The primary goal of this study is to characterize the safety, tolerability, and maximum tolerated dose (MTD) of MGD007 when combined with MGA012. Pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD), and the anti-tumor activity of the combination of MGD007 and MGA012 will also be assessed.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1b/2, dose escalation and cohort expansion study designed to characterize the safety, tolerability, PK, PD, immunogenicity, and preliminary antitumor activity of MGD007 and MGA012, administered in combination by IV infusion, in patients with histologically proven, relapsed/refractory metastatic colorectal carcinoma, irrespective of the KRAS and MMR status of their tumors.

The study consists of a Dose Escalation Phase to determine the MTD or Maximum Administered Dose (MAD; if no MTD is defined) of the combination, followed by a Cohort Expansion Phase to further define the safety and initial antitumor activity of the combination with the doses established in the Dose Escalation Phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, relapsed/refractory metastatic colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable disease per RECIST 1.1 criteria
* Participants in the Dose Escalation Phase must have had recurrence, progression or intolerance to standard therapy consisting of at least 2 prior standard regimens (containing a fluoropyrimidine plus a platinum analogue and/or irinotecan) for metastatic disease. Participants in the Cohort Expansion portion will be allowed to participate after 1 prior standard regimen. Those who are inappropriate candidates for or have refused treatment with these regimens are also eligible. No more than 5 prior therapies are permitted. Patients previously treated with MGD007 on Study Protocol CP-MGD007-01 and who did not develop antibodies to MGD007 while on the CP-MGD007-01 study, may be enrolled. Patients that were previously treated on CP-MGD007-01 will only be treated on this study once MTD/MAD has been defined.
* Availability of sufficient tumor specimens to enable retrospective determination of gpA33, CD3, PD-1, and PD-L1 expression
* 30 participants in the Cohort Expansion portion must have lesions that are accessible for paired biopsies with acceptable clinical risk in the judgment of the investigator.

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases. No concurrent treatment for the CNS disease; no progression of CNS metastases on MRI or CT for at least 14 days after last day of prior therapy for the CNS metastases; no concurrent leptomeningeal disease or cord compression
* History of known or suspected autoimmune disease with certain exceptions
* History of prior allogeneic bone marrow, stem-cell, or solid organ transplantation.
* Major surgery, systemic anti-neoplastic therapy, or investigational therapy within 4 weeks
* Radiation therapy within 2 weeks
* Systemic corticosteroids (≥ 10 mg per day prednisone or equivalent) or other immune suppressive drugs within the 14 days
* History of Grade 3 or greater drug-related diarrhea/colitis during treatment with checkpoint inhibitors including anti-LAG-3, anti-PD-1, anti PD-L1, or anti-CTLA-4 antibodies
* Clinically significant cardiovascular disease; gastrointestinal disorders; pulmonary compromise; viral, bacterial, or systemic fungal infections
* History of positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome
* History of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale School of Medicine, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 6 academic/oncology centers experienced in the conduct of clinical trials.
Groups:
- Dose Level 1: 0.4 mcg/kg MGD007 administered by intravenous (IV) infusion once per week in 8-week cycles, plus 3 mg/kg MGA012 administered by IV infusion once every 2 weeks.
- Dose Level 2: 0.6 mcg/kg MGD007 administered by intravenous (IV) infusion once per week in 8-week cycles, plus 3 mg/kg MGA012 administered by IV infusion once every 2 weeks.
- Dose Level 3: 0.8 mcg/kg MGD007 administered by intravenous (IV) infusion once per week in 8-week cycles, plus 3 mg/kg MGA012 administered by IV infusion once every 2 weeks.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 5 | 3 | 28
Safety Population | 5 (At least 1 dose of study drug) | 3 | 28
Response Evaluable Population | 5 (All patients who received at least one dose of any study drug, had baseline measurable disease, and had at least one post-baseline radiographic tumor assessment or discontinued treatment due to clearly documented, clinically progressive disease or death.) | 3 | 24
Completed | 0 | 0 | 2
Not Completed | 5 | 3 | 26
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 4 | 0 | 14
Not completed — Study Terminated | 1 | 3 | 11

BASELINE CHARACTERISTICS:
Population: Safety analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 5 | 3 | 28 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (5.13) | 46.3 (2.89) | 55.5 (7.54) | 54.5 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 13 | 16
  Male | 2 | 3 | 15 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 5 | 2 | 25 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 28 | 36
ECOG Performance Status [Count of Participants; unit: Participants]
  ECOG Performance Status 0 (Fully active without restriction) | 2 | 1 | 15 | 18
  ECOG Performance Status 1 (restricted in physically strenuous activity, but ambulatory) | 3 | 2 | 13 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse Events, Serious Adverse Events
Time Frame: Up to approximately 12 weeks
Population: All patients who received at least one dose of study drug and reporting at least one adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 5 | 3 | 28
Participants | 5 | 3 | 28

2. Secondary Outcome: Peak Plasma Concentration
Description: PK of MGD007 and MGA012 in combination
Time Frame: 7 weeks
Population: PK assays were not performed since the Sponsor has decided not to continue clinical development of MGD007.
Arm/Group | MGD007 + MGA012
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants That Develop Anti-drug Antibodies
Description: Proportion of patients who develop anti-MGD007/MGA012 antibodies, immunogenicity
Time Frame: 1 year
Population: ADA assays were not performed since the Sponsor has decided not to continue clinical development of MGD007.
Arm/Group | MGD007 + MGA012
Number analyzed (Participants) | 0

4. Secondary Outcome: The Number of Participants With Response Based on the Change in Tumor Volume
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and immune related RECIST criteria: number of patients with either complete response (CR) or partial response (PR) will determine the Overall Response Rate (ORR)
Time Frame: Every 8 weeks
Population: Response evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 5 | 3 | 24
Participants
  Stable Disease | 0 | 1 | 10
  Progressive Disease | 5 | 2 | 14

ADVERSE EVENTS:
Time Frame: Study Day 1 through study completion, average 36 days.
Description: Treatment-emergent AEs were summarized by system organ class (SOC) and preferred term (PT), by relationship to study drugs, and by highest severity. For laboratory tests, number and percent of patients shifted from baseline to post-baseline maximum severity in CTCAE grade were summarized.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/3 | 14/28
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3 | 14/28
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=5) | Dose Level 2 (N=3) | Dose Level 3 (N=28)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=5) | Dose Level 2 (N=3) | Dose Level 3 (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 7 (7)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 24 (24)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 23 (23)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2) | 16 (16)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 20 (20)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 16 (16)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 10 (10)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 7 (7)
Chills (General disorders) | 0 (0) | 0 (0) | 6 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (General disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 7 (7)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 5 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phophatase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood fibrogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 8 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Arthraligia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 5 (5)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall allow SPONSOR at least 45 days to review manuscript and at least 21 days to review poster, abstract or other material. SPONSOR can review publications solely for identifying Proprietary Information, which shall be removed upon SPONSOR's request to the extent deletion does not preclude complete/accurate presentation and interpretation of Study results; to identify patentable Inventions, and provide other comments, provided that Investigator isn't obligated to address comments.

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03531632/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT03531632/SAP_001.pdf